CLINICAL TRIAL: NCT06673329
Title: Safety and Efficacy of Brodalumab in the Treatment of Immune-Related Adverse Events: A Pilot Study
Brief Title: Brodalumab in the Treatment of Immune-Related Adverse Events
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Brian Henick, MD (Other)
Collaborators: Bausch Health (Unknown)
Responsible Party: Sponsor-Investigator, Brian Henick, MD, Assistant Professor of Medicine, Division of Hematology/Oncology, Columbia University
Organization: Columbia University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AAAV1382
Record Dates: First submitted 2024-10-31; First posted 2024-11-04 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Breast Cancer; Esophageal Cancer; Kidney Cancer; Lung Cancer; Thyroid Cancer; Gynecologic Cancer; Pancreatic Cancer; Stomach Cancer; Brain Tumor; Colon Cancer; Rectal Cancer; Head and Neck Cancer; Oral Cancer; Liver Cancer; Skin Cancer; Prostate Cancer; Testicular Cancer; Solid Tumor
MeSH Terms: conditions — Breast Neoplasms; Esophageal Neoplasms; Kidney Neoplasms; Lung Neoplasms; Thyroid Neoplasms; Pancreatic Neoplasms; Stomach Neoplasms; Brain Neoplasms; Colonic Neoplasms; Rectal Neoplasms; Head and Neck Neoplasms; Mouth Neoplasms; Liver Neoplasms; Skin Neoplasms; Prostatic Neoplasms; Testicular Neoplasms | interventions — brodalumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- brodalumab to treat irAEs in patient with solid tumors (Experimental): Brodalumab 210 mg subcutaneous injection on weeks 0, 1, 2 followed by administration every 2 weeks until week 24
  Interventions: Drug: Brodalumab; Radiation: CT scan

INTERVENTIONS:
Drug: Brodalumab — Brodalumab 210 mg subcutaneous injection
  Other Names: SILIQ
Radiation: CT scan — CT scans within 4 weeks of starting brodalumab and every 3 months during the study for tumor assessment

SUMMARY:
The purpose of this study is to test the safety and effectiveness of using brodalumab in patients who develop side effects from cancer immune therapy. Immune-related side effects are due to activation of the immune system in patients who previously received immunotherapy and the goal of this study is to help better control these side effects. Brodalumab is often used to treat patients with autoimmune diseases (diseases where the immune system is activated against normal organs) and safe doses and treatment schedules have been determined in these patients. Immune-related side effects appear to closely mirror these autoimmune conditions. Brodalumab has not been approved by the United States Food and Drug Administration (FDA) for use in immunotherapy side effects but it has been approved for treatment of autoimmune conditions.

DETAILED DESCRIPTION:
The proposed study will evaluate the safety and efficacy of brodalumab in improving and resolving Immune-Related Adverse Events (irAEs) in patients treated with brodalumab. Eligible subjects must have an immune-related adverse event with the intent to treat it with steroids. Subjects will receive subcutaneous brodalumab for 24 weeks. Peripheral blood will be collected at all in-person study visits for mechanistic studies. Participants will be evaluated at week 0, 1, 2, 4, and then every 4 weeks after that until week 24 as dictated by the standard of care using a combination of telemedicine and face-to-face evaluations. Additional safety follow-up visits will occur at weeks 28 and 36. All patients will have the Columbia Suicide Severity Rating Scale (C-SSRS), and Patient Health Questionnaire-9 (PHQ-9) administered at all visits. The treatment protocol consists of subcutaneous brodalumab 210 mg administered at baseline and then at weeks 0, 1, and 2, then bi-weekly for a total of 24 weeks (the current FDA-approved dosing for plaque psoriasis). Glucocorticoids may be used at baseline at the discretion of the investigators, with the goal of tapering off of steroids over 4-8 weeks if tolerated (see proposed taper in appendix). Continued treatment beyond the 24-week course can be evaluated by the treating investigator and the Sponsor-Investigator, weighing risks versus clinical benefit.

ELIGIBILITY:
Inclusion Criteria:

* Ability to provide written informed consent by subject or guardian
* Individuals >18 years of age
* Diagnosis of an irAE clinically suspected to be IL-17 mediated
* Intent-to-treat or prior treatment with systemic steroids for irAE management
* Histology-proven primary advanced or metastatic solid organ malignancy treated with immunotherapy. Patients being treated with curative intent are not eligible to enroll.
* Subject has a negative test for tuberculosis during screening defined as either: negative purified protein derivative (PPD) (< 5 mm of induration at 48 to 72 hours after test is placed) OR negative QuantiFERON test. Tuberculosis testing must be performed within 30 days prior to trial initiation.
* Subjects with a positive PPD and a history of Bacillus Calmette-Guérin vaccination are allowed with a negative QuantiFERON test.
* Subjects with a positive PPD test (without a history of Bacillus Calmette-Guérin vaccination) or subjects with a positive or indeterminate QuantiFERON test are allowed if they have all of the following: no symptoms of tuberculosis (defined as fever, shortness of breath, cough or night sweats), documented history of a completed course of adequate prophylaxis (per local standard of care), no known exposure to a case of active tuberculosis after most recent prophylaxis, no evidence of active tuberculosis on chest radiograph within 3 months prior to the first dose of brodalumab.

Exclusion Criteria:

* Estimated creatinine clearance < 40 mg/min
* Active suicidal ideation or severe depression (as defined by the Diagnostic and Statistical Manual of Mental Disorders Version IV criteria (DSM-IV)) at the time of enrollment or a PHQ-9 score > 20
* History of prior suicide attempts
* PHQ-9 score greater >5 and < 20 without an established mental health provider who verifies stability in their depression
* Current or prior drug or alcohol abuse within the past 6 months (as defined by the DSM IV)
* In the opinion of the investigator, the patient requires additional immunosuppressive treatment (other than corticosteroids and brodalumab)
* Known hypersensitivity or contraindication to brodalumab, corticosteroids or any components of brodalumab
* Prior treatment with brodalumab
* Pregnancy, breastfeeding, or use of a nonreliable method of contraception

  * For patients assigned female at birth: lack of willingness to use highly effective methods of birth control during treatment and for at least 4 weeks after the last dose of brodalumab (except if surgically sterile or at least 2 years postmenopausal, with postmenopausal status confirmed by Follicle-Stimulating Hormone (FSH) in the postmenopausal range).
  * Highly effective methods of birth control include: use of hormonal contraceptives that inhibit ovulation, hormone-releasing intrauterine devices, and copper intrauterine devices. Oral contraceptive pills must be supplemented by a barrier method.
  * Patients planning to become pregnant while enrolled in the study and within 4 weeks after the last dose of brodalumab will not be permitted to enroll
* Chronic or current severe infection requiring IV therapy
* Evidence of active hepatitis B, C, or tuberculosis.
* History of latent tuberculosis infection which is incompletely treated based upon local standard of care or which was never treated
* History of or active Crohn's disease.
* Myocardial infarction, unstable angina pectoris or stroke within the past 12 months prior to the first investigational product dose
* Any concurrent medical condition or electrocardiogram (ECG) abnormality that, in the opinion of the investigator, could cause this study to be detrimental to the subject.
* Any medical condition or treatment for a condition that, in the opinion of the investigator, might interfere with participation in the study or affect the reliability of clinician assessment or patient self-report
* Other known clinically significant active medical conditions, such as:

  * Severe cardiovascular disease, including advanced heart failure (American Heart Association Stage D)
  * Aspartate aminotransferase (AST) and or alanine aminotransferase (ALT) greater than 2 times the upper limit of normal or greater than 3 times the upper limit of normal in patients with liver metastases measured on at least two separate occasions
  * Direct bilirubin greater than or equal to 1.5 mg/dL in patients with or without liver metastases
  * Bone marrow insufficiency unrelated to the irAE (according to investigator judgment) with White Blood Cell (WBC) <2000/mm3, absolute neutrophil count <1500/ mm3, thrombocytopenia (platelet count) <50,000/mm3, hemoglobin < 8.0 g/dL
* Plan to proceed with further curative intent treatment for cancer at the time of enrollment despite the presence of irAE
* Participation in another therapeutic clinical trial and receipt of investigational drugs within 4 weeks before the screening visit
* Previous diagnosis of an autoimmune disease or administration of immunosuppressants in a time frame that would impede interpretation of brodalumab administration
* Planned use of immunosuppressive agents other than steroids (including infliximab, vedolizumab, tocilizumab etc.) or administration of such agents within 28 days of trial initiation
* Administration of live-virus vaccines within 4 weeks before the first dose of brodalumab

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Estimated)
Dates: Start 2025-03-11 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Number of Adverse Events | Up to 36 weeks
  The number of adverse events of each grade that occur and the number of adverse events attributed to brodalumab, as per the Common Terminology Criteria for Adverse Events version 5 (CTCAE v5).
Percentage of primary Immune-Related Adverse Event (irAE) severity decreased | 24 weeks
  The percentage of patients whose primary irAE severity decreased by >1 grade per CTCAE criteria from study completion to treatment discontinuation.

SECONDARY OUTCOMES:
Percentage net decrease in the average steroid dose required for irAE management | Up to 36 weeks
  The percentage of patients with a net decrease in the average steroid dose required for irAE management (defined by the ratio of the average steroid dose in prednisone equivalents over the 7 days following enrollment compared to the average dose in the 7 days prior to study completion).
Proportion of Patients Successfully Tapered Off Steroids | Up to 36 weeks
  The proportion of patients who can be tapered completely off of steroids (and remain off for a minimum of 1 week).
Mean Time to Complete Resolution of irAE Symptoms | Up to 36 weeks
  Mean time to complete resolution of irAE clinical manifestation ((as defined as absence of signs/symptoms consistent with the irAE or return to baseline symptoms prior to irAE development)).
Change in Tumor Burden Assessed by RECIST Criteria at 24 Weeks | 24 weeks
  Change in tumor burden as measured by RECIST criteria comparing CT/MRI scan at the time of enrollment to CT/MRI scan at 24 weeks.
Proportion of Patients with Grade 3 or Higher Infection Events | Up to 36 weeks
  The proportion of patients with > grade 3 infection per CTCAE.
Cumulative Steroid Exposure over 24 Weeks | 24 weeks
  Cumulative steroid exposure (in prednisone equivalents) over 24 weeks
FACT-G global assessment score | Baseline and 24 weeks
  Change in the quality of life as measured by the Functional Assessment of Cancer Therapy - General (FACT-G) global assessment score. Score range is 0-108. Higher scores indicate a better quality of life, while lower scores suggest worse outcomes.
Progression-free survival (PFS) | Up to 36 weeks
  PFS is defined as the duration of time from the start of treatment to the time of progression or death, whichever occurs first, measured in months
Overall Survival (OS) | Up to 36 weeks
  OS is defined as the duration of time from either the date of diagnosis or the start of treatment that patients diagnosed with the disease are still alive, measured in months.

CONTACTS AND LOCATIONS:
Overall Officials: Brian Henick, MD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Irving Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Description Herbert Irving Comprehensive Cancer Center (HICCC) Clinical Trials page — https://www.cancer.columbia.edu/